CLINICAL TRIAL: NCT06869681
Title: Comparison of Efficacy of Sertaconazole Nitrate Cream 2 Percent Vs Clotrimazole 1 Percent for the Treatment of Tinea Pedis.
Brief Title: Efficacy of Tropical Sertaconazole Nitrate 2% Vs Clotrimazole 1% for Tinea Pedis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Dr. Madhoo, MBBS, Doctor, FCPS Trainee, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No.F.2-81/2024-GENL/88/JPMC; No.F.2-81/2024-GENL/88/JPMC (Other: Jinnah Postgraduate Medical Centre(JPMC))
Record Dates: First submitted 2025-02-25; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Tinea Pedis
Keywords: Tinea Pedis; Efficacy; Sertaconazole Nitrate Cream; Clotrimazole
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group-A topical Sertaconazole 2% (Experimental): After cleaning the identified lesions, the patients will topically self-apply the topical Sertaconazole 2% creams using a cotton swab applicator, where the applied amount will be able to make the lesions be covered with a thin layer of medication. The creams will be applied topically twice daily for 4 weeks.
  Patients will be followed up weekly for clinical improvement and side-effects of therapy upto 4 weeks of the treatment.
  Interventions: Drug: Topical Sertaconazole 2%
- Group-B Clotrimazole 1% (Experimental): After cleaning the identified lesions, the patients will topically self-apply the Clotrimazole 1% creams using a cotton swab applicator, where the applied amount will be able to make the lesions be covered with a thin layer of medication. Both the creams will be applied topically twice daily for 4 weeks.
  Interventions: Drug: Clotrimazole 1%

INTERVENTIONS:
Drug: Topical Sertaconazole 2% — After cleaning the identified lesions, the patients will topically self-apply the both products/creams using a cotton swab applicator, where the applied amount will be able to make the lesions be covered with a thin layer of medication. Both the creams will be applied topically twice daily for 4 weeks.
  Arms: Group-A topical Sertaconazole 2%
Drug: Clotrimazole 1% — Same as above
  Arms: Group-B Clotrimazole 1%

SUMMARY:
This randomized controlled trail study will be carried out on OPD patients in the Department of Dermatology, Jinnah Postgraduate Medical Center. Institutional Ethical committee permission will be obtained and clinical trial registration number (CTN) will be obtained for the study. Written consent will obtained from all the participants of the study.

All the diagnosed patients of Tinea Pedis who will meet the selection criteria will be enrolled and will be educated regarding the study. Participants will be randomly allocated in into two groups utilizing envelop method; patients of Group-A will use topical Sertaconazole 2% and patients in Group-B will use Clotrimazole 1%.

Randomization: Random number sequence will be generated on computer by a simple randomization schedule. Each randomization number will be sealed in an opaque envelope with a serial number on it. The patient with a known serial number opened the corresponding envelope to be informed of the assignment.

Treatment: After cleaning the identified lesions, the patients will topically self-apply the both products/creams using a cotton swab applicator, where the applied amount will be able to make the lesions be covered with a thin layer of medication. Both the creams will be applied topically twice daily for 4 weeks.

Patients will be followed up weekly for clinical improvement and side-effects of therapy upto 4 weeks of the treatment. At final follow up (after 4 week of treatment), the patients will be evaluated by all clinical investigations and microscopic examination (10% potassium hydroxide) of a skin scraping from site of the lesion. Adverse effects of the drugs among all patients will also be recorded. The photograph of the lesions taken before treatment and at the end of the study will be used for assessing the clinical improvement of the cases.

Detailed questionnaires will be followed regarding demographic and clinical characteristics like age, BMI, symptoms and co morbidities etc. Proper selection criteria will be used to control any biasness. Efficacy will be reported as per operational definition. In case of, topical therapy will be terminated and the concerned patient will be switched over to an oral antifungal drug at the discretion of the dermatologist. Any adverse events during the study will also be reported.

DETAILED DESCRIPTION:
This randomized controlled trail study will be carried out on OPD patients in the Department of Dermatology, Jinnah Postgraduate Medical Center. Institutional Ethical committee permission will be obtained and clinical trial registration number (CTN) will be obtained for the study. Written consent will obtained from all the participants of the study.

All the diagnosed patients of Tinea Pedis who will meet the selection criteria will be enrolled and will be educated regarding the study. Participants will be randomly allocated in into two groups utilizing envelop method; patients of Group-A will use topical Sertaconazole 2% and patients in Group-B will use Clotrimazole 1%.

Randomization: Random number sequence will be generated on computer by a simple randomization schedule. Each randomization number will be sealed in an opaque envelope with a serial number on it. The patient with a known serial number opened the corresponding envelope to be informed of the assignment.

Treatment: After cleaning the identified lesions, the patients will topically self-apply the both products/creams using a cotton swab applicator, where the applied amount will be able to make the lesions be covered with a thin layer of medication. Both the creams will be applied topically twice daily for 4 weeks.

Patients will be followed up weekly for clinical improvement and side-effects of therapy upto 4 weeks of the treatment. At final follow up (after 4 week of treatment), the patients will be evaluated by all clinical investigations and microscopic examination (10% potassium hydroxide) of a skin scraping from site of the lesion. Adverse effects of the drugs among all patients will also be recorded. The photograph of the lesions taken before treatment and at the end of the study will be used for assessing the clinical improvement of the cases.

Detailed questionnaires will be followed regarding demographic and clinical characteristics like age, BMI, symptoms and co morbidities etc. Proper selection criteria will be used to control any biasness. Efficacy will be reported as per operational definition. In case of, topical therapy will be terminated and the concerned patient will be switched over to an oral antifungal drug at the discretion of the dermatologist. Any adverse events during the study will also be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 18-65 years age.
* Either sex.
* Patients presenting with the clinical manifestations of tinea pedis such as erythema, scaling, vesicles, pustules, and itch.
* Skin scrapings positive for KOH mount test.

Exclusion Criteria:

* Patients with secondary bacterial infection.
* Patients using topical or taken any oral antifungal drug before the baseline visit.
* Diabetic, immunocompromised patients.
* Women with pregnancy or lactating mothers.
* Patients allergic to the drugs in this study.
* Those who withdrew in the middle of the study, or changed drugs without authorization will also be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
frequency of Efficacy in both treatment groups | 4 weeks
  Reduction in total composite score of at least 2 points with negative KOH test after 4 week of treatment and reporting of no adverse events will be considered as efficacy of the treatments

IPD SHARING:
Plan to Share IPD: No